CLINICAL TRIAL: NCT05210868
Title: A Phase I/II Open-Label, Single-Arm, Multicenter Clinical Study of CM355 in Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma (B-NHL)
Brief Title: A Phase I/II Study of CM355 in Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma (B-NHL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM355-001
Record Dates: First submitted 2021-12-09; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-11

CONDITIONS: Hematoma
MeSH Terms: conditions — Hematoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM355 (Experimental): 1. Dose Escalation Phase CM355
  2. Dose Expansion Phase CM355
  Interventions: Drug: CM355

INTERVENTIONS:
Drug: CM355 — 1. Dose Escalation Phase CM355 will be taken by patients and will be treated follow the "3+3" dose escalation scheme
  2. Expansion Phase CM355 will be taken by patients and will assess the efficacy of CM355 in patients with specific histopathological Non-Hodgkin's Lymphoma, and the safety of drug

SUMMARY:
A Phase I/II Open-Label, Single-Arm, Multicenter Clinical Study of CM355 in Patients With R/R B-NHL

DETAILED DESCRIPTION:
This is a phase I/II open-label, single-arm, multicenter study in China to evaluate the safety, tolerability, and efficacy of CM355 in patients with R/R B-NHL. In the study, patients will not be screened for CD20 expression, but they must have a diagnosis of B-NHL that is expected to express CD20. After enrollment, tumor samples will be collected for retrospective analysis of CD20 expression

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years old.
2. Eastern Cooperative Oncology Group (ECOG, see Appendix 3) PS score of 0-1.
3. Histopathologically confirmed relapsed or refractory B-cell NHL has been confirmed or anticipated to express CD20 in lymphoma lesions.
4. According to Lugano criteria, imaging evaluation shows at least one bidimensionally measurable lesion.
5. The level of organ function of patients must In line with the testing standard of the clinical trial center prior to the first dose of the investigational drug
6. Expected survival ≥ 3 months.
7. All toxicities caused by prior anticancer therapy must have recovered to grade ≤ 1 (based on CTCAE v5.0) except alopecia and fatigue.
8. Female patients with childbearing potential should have a negative blood pregnancy test result within 7 days prior to the first dose.
9. Female patients with childbearing potential or male patients and their partners must agree to take effective contraceptive measures from the signing of the ICF to at least 6 months after the last dose of investigational drug.
10. Female patients cannot breastfeed or plan to become pregnant during the study until at least 6 months after the last dose of investigational drug.
11. The patient voluntarily joined the study and signed the ICF.

Exclusion Criteria:

1. Active or past central nervous system (CNS) lymphoma.
2. Other active malignancies occurring within 5 years prior to the first dose of investigational drug, with the exception of radically treated local curable cancers.
3. The patient has a disease or medical history that needs to be excluded as specified in the Clinical Trial Protocol.
4. Any active infection requiring systemic therapy via intravenous infusion within 14 days prior to the first dose of investigational drug.
5. According to the trial scheme, patients infected with hepatitis B virus, hepatitis C virus, HIV, EBV, CMV, syphilis, or patients with active pulmonary tuberculosis or history of pulmonary tuberculosis infection are not suitable to participate in the study.
6. Any severe or uncontrolled systemic disease.
7. History of severe allergic reactions (CTCAE v5.0 classification is greater than 3 grades) to humanized monoclonal antibodies, or known hypersensitivity to any component of CM355.
8. Any mental or cognitive disorder that may limit the patient's understanding and execution of the ICF and compliance with the study.

   Medication history and surgical history:
9. Having received allogeneic hematopoietic stem cell transplantation or received auto-HSCT within 100 days prior to the first dose.
10. Active bleeding within 2 months prior to screening, or receiving anticoagulants, or other bleeding symptoms requiring medical intervention.
11. Having undergone major surgery within 28 days prior to the first dose, or minor surgery within 2 weeks prior to the first dose; invasive examinations for the purpose of diagnosis are not considered as surgery; except for the insertion of vascular access device.
12. Patients who experienced grade ≥ 3, severe or life-threatening immune-related adverse events or grade 1-2 immune-related adverse events that did not return to baseline levels after treatment discontinuation in a previous immunotherapy.
13. Patients who have received any other investigational anti-cancer drug therapy within 28 days prior to the first dose.
14. Inoculation of live attenuated vaccines within 28 days prior to the first dose, or anticipation that live attenuated vaccines will be required during the study.
15. Patients who have received any drugs therapy that need to be excluded from the Clinical Trial Protocol within a certain period of time for the first administration.
16. Prior participation in other clinical trials within 28 days prior to the first dose of the investigational drug, or planning to participate in this study and other clinical trials at the same time.
17. Known alcoholism or drug abuse history.
18. Other conditions determined by the investigator that render patients unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | Up to 2 year
  Incidence, nature, and severity of dose-limiting toxicities.
Recommended phase II dose (RP2D) and/or (maximum tolerated dose) MTD | Up to 2 year
  To determine the recommended phase II dose (RP2D) and/or the maximum tolerated dose (MTD) of CM355 in patients with R/R B-NHL.
Objective response rate（ORR） | through study completion，an average of 5 year
  Objective response rate (ORR) as assessed by independent review committee (IRC)
The safety and tolerability of CM355 | through study completion，an average of 5 year
  Incidence, nature, and severity of adverse events (AEs) as judged according to NCI-CTCAE v5.0.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Every cycle (21 days), until the end of treatment
  Dose Escalation peak plasma concentration (ng/mL)
Area under the plasma concentration versus time curve (AUC) | Every cycle (21 days), until the end of treatment
  Dose Escalation AUC（μg·h/mL）
Peak time | Every cycle (21 days), until the end of treatment
  Time of maximum observed plasma concentration (Tmax)
T1/2 | Every cycle (21 days), until the end of treatment
  Terminal half-life of CM355
Clearanc (CL) | Every cycle (21 days), until the end of treatment
  Total body clearance of the drug from plasma (CL) of CM355
Anti-CM355 antibodies (ADAs) | Every cycle (21 days), until the end of treatment
  Incidence of anti-CM355 antibodies (ADAs) and their correlation with clinical outcomes.
Objective response rate (ORR) | through study completion，an average of 5 year
  Objective response rate (ORR) as assessed by investigators
Complete response rate (CRR) | through study completion，an average of 5 year
  Complete response rate (CRR) as assessed by investigators or independent review committee (IRC)
Duration of response (DOR) | through study completion，an average of 5 year
  Duration of response (DOR) as assessed by investigators or Independent review committee (IRC)
Progression-Free-Survival (PFS) | through study completion，an average of 5 year
  Progression-Free-Survival (PFS) as assessed by investigators or independent review committee (IRC)
overall survival (OS) | through study completion，an average of 5 year
  overall survival (OS) as assessed by investigators or independent review committee (IRC)

OTHER OUTCOMES:
Cytokines | Up to 17 cycles （21 days per cycle)
  To conduct qualitative and quantitative analyses of the level of changes in cytokines (IL-2, IL-6, IL-10, INF-γ, and TNF-α).

CONTACTS AND LOCATIONS:
Overall Officials: Yuqin Song, M.D., Principal Investigator — Beijing university cancer hospital
Locations (1):
- Beijing university cancer hospital, Beijing, China